CLINICAL TRIAL: NCT07101094
Title: Real-world Evaluation of Treatment Satisfaction and KarXT Utilization Registry (RESKU)
Brief Title: Evaluation of Treatment Satisfaction and KarXT Utilization Registry (RESKU)
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CN012-0066
Record Dates: First submitted 2025-07-23; First posted 2025-08-03 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — xanomeline; trospium chloride; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants receiving xanomeline and trospium chloride (X/T) therapy
  Interventions: Drug: xanomeline and trospium chloride (X/T) therapy

INTERVENTIONS:
Drug: xanomeline and trospium chloride (X/T) therapy — According to the product label

SUMMARY:
The purpose of this study is to understand treatment preference and satisfaction among adults with schizophrenia in the United States who are prescribed xanomeline and trospium chloride (X/T) therapy

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years at index date.
* Have a confirmed diagnosis of schizophrenia before index date.
* Receipt of an initial prescription order for xanomeline and trospium chloride (XT) and plan to fill and initiate such therapy.
* Provide a signed and dated Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved written informed consent form (ICF) in accordance with regulatory, local, and institutional guidelines.
* Agree to use an electronic device to record, or provide paper entry of, patient-reported outcomes (in English or Spanish).
* English or Spanish speaking.

Exclusion Criteria:

* Participation in an interventional study within the last 30 days or plan to participate in such study at the time of eligibility screening.
* Evidence of use of XT prior to time of eligibility screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adults diagnosed with schizophrenia who initiate treatment with xanomeline and trospium chloride (XT) in the US.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-05-14 (Estimated)

PRIMARY OUTCOMES:
Participant medication preference as assessed by the Preference of Medication (POM) questionnaire | Month 1, Month 3, Month 6
Participant treatment satisfaction as assessed by the Medication Satisfaction Questionnaire (MSQ) | Baseline, Month 1, Month 3, Month 6

SECONDARY OUTCOMES:
Treatment titration plan as described by the treating clinician | Baseline, Month 1, Month 3, Month 6
Treatment switch plan as described by the treating physician | Baseline, Month 1, Month 3, Month 6
Treatment dose prescribed | Baseline, Month 1, Month 3, Month 6
Concomitant medication prescribed | Baseline, Month 1, Month 3, Month 6
Number of participants who are prescribed a treatment dose change | Month 1, Month 3, Month 6
Reasons for treatment discontinuation | Month 1, Month 3, Month 6
Participant baseline clinical characteristics | Baseline
Participant baseline demographics | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (16):
- United States (16):
  - Local Institution - 0009, Orange, California
  - Local Institution - 0010, San Jose, California
  - Local Institution - 0003, Evanston, Illinois
  - Local Institution - 0007, Baltimore, Maryland
  - Local Institution - 0004, Catonsville, Maryland
  - Local Institution - 0008, Belmont, Massachusetts
  - Local Institution - 0002, Boston, Massachusetts
  - Mayflower Clinical, South Dartmouth, Massachusetts
  - Omaha Insomnia and Psychiatric Services, Omaha, Nebraska
  - Hackensack Meridian Health - Carrier Clinic, Belle Mead, New Jersey
  - Local Institution - 0015, New York, New York
  - Local Institution - 0016, Kinston, North Carolina
  - Local Institution - 0014, Westlake, Ohio
  - Continuum Health Providers, Fort Mill, South Carolina
  - Local Institution - 0012, El Paso, Texas
  - Local Institution - 0013, Longview, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts